CLINICAL TRIAL: NCT07118943
Title: A Clinical Study to Determine the Efficacy of Four Test Articles to Improve Skin Longevity Over Eight Weeks Use Period
Brief Title: Efficacy of Four Topical Products to Improve Skin Longevity
Acronym: Before/After
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amazentis SA (Industry)
Collaborators: Princeton Consumer Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ASACLI1W
Record Dates: First submitted 2025-08-04; First posted 2025-08-12 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Aging; Wrinkle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Face care product (eye cream) (Experimental): The topical product (eye cream) containing Mitopure will be used for eight weeks.
  Interventions: Other: Face care product
- Face care product (cream A) (Experimental): The topical product (moisturizing formula A) containing Mitopure will be used for eight weeks.
  Interventions: Other: Face care product
- Face care product (cream B) (Experimental): The topical product (moisturizing formula B) containing Mitopure will be used for eight weeks.
  Interventions: Other: Face care product
- Face care product (serum) (Experimental): The topical product (serum) containing Mitopure will be used for eight weeks.
  Interventions: Other: Face care product

INTERVENTIONS:
Other: Face care product — The topical product will be applied twice daily (morning and night).
  Arms: Face care product (cream A)
Other: Face care product — The topical product will be applied twice daily (morning and night).
  Arms: Face care product (cream B)
Other: Face care product — The topical product will be applied twice daily (morning and night).
  Arms: Face care product (eye cream)
Other: Face care product — The topical product will be applied twice daily (morning and night).
  Arms: Face care product (serum)

SUMMARY:
The objective of this study is to determine the efficacy of four topical products to improve facial skin longevity over an eight-week use period utilizing analysis of images and self-perception questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female and male volunteers aged 40 to 65 years with no signs of skin disorders.
* Subject is willing and able to read, understand, and provide written Informed Consent and signed photo release.
* Subject has a score of 3.0 to 6.0 for clinically graded visible facial wrinkles using the Fitzpatrick Classification of Facial Wrinkling scale at Baseline, to determine eligibility for the creams or serum test articles or 3.0 to 6.0 for clinically graded visible wrinkles in the eye area using a wrinkling scale for the eye cream test article.
* Subject is willing to refrain from applying/using moisturizer, creams, serums or treatment/anti-aging products to their face during the three days prior to Visit 1 (Baseline). Subject's other regular skin products such as cleanser, sunscreen and cosmetics are acceptable.
* Subject is willing to come to the test facility with a clean face free of makeup and sunscreen prior to all visits.
* Subject is a regular sunscreen user (uses at least 2 times a week).
* Subject is willing to avoid direct sun exposure and/or to apply sunscreen to their face in the event of sun exposure.
* Subject agrees to remove jewelry and false eye lashes before the visits.
* Subject agrees not to introduce any new personal care products or cosmetics to the face while participating on the study.
* Subject is willing to avoid use of tanning beds and any use of sunless tanners on the face throughout the study.
* Subject is willing to follow study instructions and available to attend all the study visits.
* Male only: Male subjects are willing to come to all visits with a clean-shaven face. Goatee and/or mustache are acceptable.

Exclusion Criteria:

* Female only: Pregnant or lactating or planning a pregnancy during the course of the study. (self-reported).
* Piercing or tattoos including permanent or semi-permanent make-up on the face which may interfere with study assessments.
* Any conditions on the face that would interfere with evaluations (i.e. full beard, scars, open cuts, sunburn, severe hyperpigmentation, facial hair/peach fuzz, etc.) or active acne or acne marks.
* Any skin conditions such as rosacea, eczema, psoriasis, seborrheic dermatitis, vitiligo, etc., or is under the treatment of a doctor for any skin condition on the face.
* Use of a self-tanner/stain on the face within two weeks of the study start.
* Allergies or sensitivities to facial moisturizer products, similar materials or their ingredients or cosmetics.
* Insulin-dependent diabetes.
* Hematological or immune deficiency disease such as HIV positive, AIDS, Systemic Lupus Erythematosus.
* Recent use within the last 14 days of a chemical peel or is currently using an in-home or professional chemical peel on their facial skin.
* Subject has had a cosmetic medical procedure in the test area such as injectable anti-wrinkle products (e.g. Botox), facial cosmetic surgery, etc. in the last year.
* Current use of OTC (over the counter) pain medication ingested in quantities exceeding label use.
* Use of topical treatments such as OTC (over-the-counter) acne medication, hydroquinone, or hydrocortisone on the face in the last month.
* Currently participating in another clinical study or trial involving the face.
* Subject has been diagnosed with any type of cancer especially skin cancer within the past 12 months or treated for cancer in the last 5 years.
* Subject has any medical condition which, in the opinion of the Investigator, would compromise the safety of the subject or confound study results.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2025-08-12 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2025-10-09 (Actual)

PRIMARY OUTCOMES:
Product Acceptance | 8 weeks
  Product Acceptance will be evaluated via questionnaire (measurement tool) responses after eight weeks of product use (time frame) and quantified as a single percentage score (unit of measure=%; minimum value=0%; maximum value=100%) so higher scores (closer to 100%) represent better Product Acceptance.
  Participants will respond to 12 closed questions by ticking one of four predefined options: -2=Fully disagree; -1=Rather disagree; 1=Rather agree; 2=Fully agree. For each question, every participant's response will be categorized as "disagree" (scores -2, -1) or "agree" (scores 1, 2). The percentage of participants that respond "agree" will be calculated ([number of "agree" responses/total number of responses]*100%), yielding one overall "agreement" value (unit of measure = %) for each of the 12 questions. Product Acceptance will be calculated by averaging the 12 overall "agreement" values. Clear product acceptance will be determined if the Product Acceptance score is at least 70%.

SECONDARY OUTCOMES:
Skin wrinkles | 8 weeks
  Three-dimensional facial images will be taken with Phaseshift Rapid In vivo Measurement Of the Skin (PRIMOS) at baseline, week 4, and week 8 and will be analyzed for skin wrinkle size (unit of measure is millimeters).
Haut AI Facial Analysis | 8 weeks
  High resolution digital facial VISIA images will be taken of right side, left side and front of the face with VISIA® CRP-GEN 5 at baseline, week 4, and week 8. The front face image will be analyzed by Haut AI for overall facial age health score (scale of 0 to 100, in which higher score represents better outcome).
Self-perceived product traits | 8 weeks
  Subjective evaluation of 12 product traits assessed via questionnaire after 4 and 8 weeks. Product traits will be assessed by the subjects with a list of closed questions with the following predefined identical options to tick: -2 = Fully disagree; -1 = Rather disagree; 1 = Rather agree; 2 = Fully agree.
  Self-perceived product trait will be calculated for each of the 12 product traits independently. For each trait, total percentages resulting in at least 80% agreement will represent a clear level of agreement and opinion of the panel. Frequencies between 70% to 80% will represent a high level of agreement. Less than 70% agreement will represent constrained and undecided agreement.
Adverse Events | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nalini Kaul, PhD, Principal Investigator — Princeton Consumer Research Corp.
Locations (1):
- Princeton Consumer Research Corp., Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No